CLINICAL TRIAL: NCT05173246
Title: JS001 Combined With Nab-paclitaxel and Cisplatin or Carboplatin as First-line Treatment for Unresectable or Advanced Small Cell Esophageal Carcinoma : a Prospective, Single Arm, Multicenter, Phase II Clinical Trial
Brief Title: JS001 Combined With TP as First-line Treatment for Unresectable or Advanced Small Cell Esophageal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other); CSPC Ouyi Pharmaceutical Co., Ltd. (Industry); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, : Professor, Principal Investigator, President, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP+JS001 in unresectable SCCE
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Small Cell Carcinoma
Keywords: JS001; Nab-paclitaxel and; Cisplatin; Carboplatin; Small cell esophageal carcinoma
MeSH Terms: interventions — Injections; 130-nm albumin-bound paclitaxel; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: JS001 Combined With TP as First-line Treatment for Unresectable or Advanced Esophageal Small Cell Carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JS001 Combined With TP (Experimental): recombinant humanized anti-PD-1 monoclonal antibody for injection (JS001) in combination with nab-paclitaxel and cisplatin or carboplatin for injection
  Interventions: Drug: JS001; Drug: nab-paclitaxel; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: JS001 — JS001 240mg, ivdrip, d1, Q3w
  Other Names: recombinant humanized anti-PD-1 monoclonal antibody for injection
Drug: nab-paclitaxel — nab-paclitaxel 220 mg/m2,ivdrip, d1,d8,Q3w
  Other Names: Paclitaxel for injection (Albumin Bound)
Drug: Cisplatin — Cisplatin 75mg/m2, ivdrip,d1,Q3w
  Other Names: Cisplatin for injection
Drug: Carboplatin — Carboplatin AUC 5,d1,Q3w
  Other Names: Carboplatin for injection

SUMMARY:
Small cell esophageal carcinoma (SCCE) is a kind of malignant tumor with poor prognosis. Our study found that the mutation spectrum and somatic CNV spectrum of SCCE were similar to those of esophageal squamous cell carcinoma (ESCC). Paclitaxel combined with cisplatin or carboplatin is the first-line treatment for ESCC. JS001 is a Chinese anti-PD-1 monoclonal antibody, which has been approved for the treatment of melanoma. This is a prospective, single arm, multicenter, phase II clinical trial of JS001 combined with nab-paclitaxel and cisplatin or carboplatin in the first-line treatment of unresectable or advanced SCCE. Aim to evaluate the safety and efficacy of this regimen in patients with unresectable or advanced SCCE.

DETAILED DESCRIPTION:
Small cell esophageal carcinoma (SCCE) is a kind of malignant tumor with poor prognosis. Our previous studies found that the mutation spectrum and somatic CNV spectrum of SCCE were similar to those of esophageal squamous cell carcinoma (ESCC). Paclitaxel combined with cisplatin or carboplatin is a common first-line treatment for ESCC. In addition, some studies have shown that PD-1 mAb combined with paclitaxel chemotherapy in esophageal cancer has better efficacy and tolerability than chemotherapy alone. JS001 is a Chinese monoclonal antibody against PD-1 for injection, which has been approved for the treatment of melanoma. This is a prospective, single arm, multicenter, phase II clinical trial of JS001 combined with nab-paclitaxel and cisplatin or carboplatin in the first-line treatment of unresectable or advanced SCCE. Aim to evaluate the safety and efficacy of this regimen in patients with unresectable or advanced SCCE.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-75 years;
2. Histologically or cytologically confirmed esophageal small cell carcinoma with unresectable locally advanced / recurrent or distant metastasis
3. Patients who have not received systemic anti-tumor therapy
4. Patients with recurrence or metastasis more than 6 months after the end of adjuvant or neoadjuvant chemotherapy accompanied by radical surgery or radical chemoradiotherapy;
5. With at least 1 measurable lesion according to RECIST 1.1 criteria;
6. ECOG score 0-1;
7. Expected survival ≥3 months;
8. Good organ function (without blood transfusion, use of hematopoietic stimulating factors, or transfusion of albumin or blood products within 7 days prior to examination): 1) Platelet (PLT) count ≥75,000 /mm3; 2) Neutrophil count (ANC) ≥1,500 /mm3; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4) Total bilirubin (TBIL) level ≤1.5×ULN; 5) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 6) Alkaline phosphatase level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 7) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance >50 ml/min;
9. Females of child bearing age must have anegative pregnancy test, and have to take contraception measures and for 3 months after the last dose
10. Able to understand and willing to sign written informed consent form.
11. Patients who agree to provide previously stored tumor tissue samples or perform biopsy to collect tumor tissue for gene testing.

Exclusion Criteria:

1. Known allergy to study drug or excipients, or allergy to similar drugs;
2. Received anti-tumor cytotoxic drug therapy, biological drug therapy (such as monoclonal antibody), immunotherapy (such as interleukin-2 or interferon) or other research drug therapy within 4 weeks before enrollment.
3. Received tyrosine kinase inhibitor treatment within 2 weeks before enrollment.
4. Patients received radiotherapy within 4 weeks or radiopharmaceuticals within 8 weeks, except for local palliative radiotherapy for bone metastases.
5. Major surgery was performed or not completely recovered from the previous surgery within 4 weeks before enrollment (the definition of major surgery refers to the level 3 and level 4 surgery specified in the administrative measures for clinical application of medical technology implemented on May 1, 2009).
6. The toxicity of previous anti-tumor therapy has not recovered to CTCAE [version 4.03] 0-1, except for the following cases: a) lipsotrichia；b) Pigmentation;c) Peripheral neurotoxicity has recovered to < CTCAE 2;d) The long-term toxicity caused by radiotherapy could not be recovered according to the judgment of the researchers;
7. Subjects with clinically symptomatic CNS metastases and/or cancerous meningitis. The subjects who have received brain or meningeal metastasis treatment in the past, if the clinical stability has been maintained for at least 2 months, and the systemic hormone treatment has been stopped for more than 4 weeks can be included.
8. Have or are currently suffering from other malignancies (except for non melanoma basal cell carcinoma of the skin, breast / cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment in the past five years).
9. Subjects have any active autoimmune disease or history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma in childhood who have completely remission and do not need any intervention in adulthood can be included; subjects with asthma requiring bronchodilator for medical intervention can not be included).
10. Previous use of anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell costimulation or checkpoint pathway).
11. Subjects with active pulmonary tuberculosis (TB) are receiving antituberculosis treatment or received antituberculosis treatment within one year before screening.
12. Patients with complications requiring long-term use of immunosuppressive drugs or systemic or local use of corticosteroids with immunosuppressive effect (dose > 10mg / day of prednisone or other therapeutic hormones).
13. Received any anti infection vaccine (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks before enrollment.
14. Pregnant or lactating women.
15. HIV positive.
16. HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 CPS / ml).
17. HCV antibody positive.
18. Researchers believe that it can affect the compliance of the protocol, or affect the subject to sign the informed consent(ICF), or any other disease or condition of clinical significance that is not suitable to participate in this clinical trial.
19. There are clinical symptoms or diseases that can not be well controlled, such as: (1) heart failure of NYHA grade 2 or above (2) unstable angina pectoris (3) myocardial infarction within one year (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Objective response rate (ORR)=CR+PR

SECONDARY OUTCOMES:
Progression free survival (PFS) | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS is the time measured from the date of initiation of treatment to the date of progression or death due to any cause, whichever occurs first.
Overall survival (OS) | from the initiation date of first cycle to the date of date of death from any cause, assessed up to 2 years
  Overall survival (OS) is the time calculated from the initiation of treatment to date of death or censored at last follow-up.
DCR | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Disease control rate (DCR) =CR+PR+SD
Six-month progression-free survival rate | from the initiation date of first cycle to six months later
  Six-month progression-free survival rate is the survival rate calculated at the end of the 6-month follow-up.
One year survival rate | from the initiation date of first cycle to one year later
  One year progression-free survival rate is the survival rate calculated at the end of the 1-year follow-up.
Severe toxicity | from the initiation date of first cycle to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nishimaki T, Suzuki T, Nakagawa S, Watanabe K, Aizawa K, Hatakeyama K. Tumor spread and outcome of treatment in primary esophageal small cell carcinoma. J Surg Oncol. 1997 Feb;64(2):130-4. doi: 10.1002/(sici)1096-9098(199702)64:23.0.co;2-c. PMID 9047250
- [Background] Hosokawa A, Shimada Y, Matsumura Y, Yamada Y, Muro K, Hamaguchi T, Igaki H, Tachimori Y, Kato H, Shirao K. Small cell carcinoma of the esophagus. Analysis of 14 cases and literature review. Hepatogastroenterology. 2005 Nov-Dec;52(66):1738-41. PMID 16334769
- [Background] Chen WW, Wang F, Chen S, Wang L, Ren C, Luo HY, Wang FH, Li YH, Zhang DS, Xu RH. Detailed analysis of prognostic factors in primary esophageal small cell carcinoma. Ann Thorac Surg. 2014 Jun;97(6):1975-81. doi: 10.1016/j.athoracsur.2014.02.037. Epub 2014 Apr 14. PMID 24726599
- [Background] Gao R, Zhang Y, Wen XP, Fu J, Zhang GJ. Chemotherapy with cisplatin or carboplatin in combination with etoposide for small-cell esophageal cancer: a systemic analysis of case series. Dis Esophagus. 2014 Nov-Dec;27(8):764-9. doi: 10.1111/dote.12149. Epub 2013 Oct 10. PMID 24118373
- [Background] Mortezaee K. Immune escape: A critical hallmark in solid tumors. Life Sci. 2020 Oct 1;258:118110. doi: 10.1016/j.lfs.2020.118110. Epub 2020 Jul 19. PMID 32698074
- [Background] Jiang X, Wang J, Deng X, Xiong F, Ge J, Xiang B, Wu X, Ma J, Zhou M, Li X, Li Y, Li G, Xiong W, Guo C, Zeng Z. Role of the tumor microenvironment in PD-L1/PD-1-mediated tumor immune escape. Mol Cancer. 2019 Jan 15;18(1):10. doi: 10.1186/s12943-018-0928-4. PMID 30646912
- [Background] Fritz JM, Lenardo MJ. Development of immune checkpoint therapy for cancer. J Exp Med. 2019 Jun 3;216(6):1244-1254. doi: 10.1084/jem.20182395. Epub 2019 May 8. PMID 31068379
- [Background] O'Donnell JS, Teng MWL, Smyth MJ. Cancer immunoediting and resistance to T cell-based immunotherapy. Nat Rev Clin Oncol. 2019 Mar;16(3):151-167. doi: 10.1038/s41571-018-0142-8. PMID 30523282
- [Background] Chen L. Co-inhibitory molecules of the B7-CD28 family in the control of T-cell immunity. Nat Rev Immunol. 2004 May;4(5):336-47. doi: 10.1038/nri1349. No abstract available. PMID 15122199
- [Background] Huang J, Mo H, Zhang W, Chen X, Qu D, Wang X, Wu D, Wang X, Lan B, Yang B, Wang P, Zhang B, Yang Q, Jiao Y, Xu B. Promising efficacy of SHR-1210, a novel anti-programmed cell death 1 antibody, in patients with advanced gastric and gastroesophageal junction cancer in China. Cancer. 2019 Mar 1;125(5):742-749. doi: 10.1002/cncr.31855. Epub 2018 Dec 3. PMID 30508306
- [Background] Mo H, Huang J, Xu J, Chen X, Wu D, Qu D, Wang X, Lan B, Wang X, Xu J, Zhang H, Chi Y, Yang Q, Xu B. Safety, anti-tumour activity, and pharmacokinetics of fixed-dose SHR-1210, an anti-PD-1 antibody in advanced solid tumours: a dose-escalation, phase 1 study. Br J Cancer. 2018 Aug;119(5):538-545. doi: 10.1038/s41416-018-0100-3. Epub 2018 May 14. PMID 29755117
- [Background] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Background] Shui L, Cheng K, Li X, Shui P, Zhou X, Li J, Yi C, Cao D. Study protocol for an open-label, single-arm, phase Ib/II study of combination of toripalimab, nab-paclitaxel, and gemcitabine as the first-line treatment for patients with unresectable pancreatic ductal adenocarcinoma. BMC Cancer. 2020 Jul 9;20(1):636. doi: 10.1186/s12885-020-07126-3. PMID 32646394
- [Background] Qiu H. Safety and efficacy of toripalimab in advanced gastric cancer: A new clinical trial bringing hope for immunotherapy in gastric cancer. Cancer Commun (Lond). 2020 Apr;40(4):194-196. doi: 10.1002/cac2.12019. Epub 2020 Apr 11. No abstract available. PMID 32277740
- [Background] Lu M, Zhang P, Zhang Y, Li Z, Gong J, Li J, Li J, Li Y, Zhang X, Lu Z, Wang X, Zhou J, Peng Z, Wang W, Feng H, Wu H, Yao S, Shen L. Efficacy, Safety, and Biomarkers of Toripalimab in Patients with Recurrent or Metastatic Neuroendocrine Neoplasms: A Multiple-Center Phase Ib Trial. Clin Cancer Res. 2020 May 15;26(10):2337-2345. doi: 10.1158/1078-0432.CCR-19-4000. Epub 2020 Feb 21. PMID 32086343
- [Background] Wang F, Liu DB, Zhao Q, Chen G, Liu XM, Wang YN, Su H, Qin YR, He YF, Zou QF, Liu YH, Lin YE, Liu ZX, Bei JX, Xu RH. The genomic landscape of small cell carcinoma of the esophagus. Cell Res. 2018 Jul;28(7):771-774. doi: 10.1038/s41422-018-0039-1. Epub 2018 May 4. No abstract available. PMID 29728688
- [Background] Antonia SJ, Lopez-Martin JA, Bendell J, Ott PA, Taylor M, Eder JP, Jager D, Pietanza MC, Le DT, de Braud F, Morse MA, Ascierto PA, Horn L, Amin A, Pillai RN, Evans J, Chau I, Bono P, Atmaca A, Sharma P, Harbison CT, Lin CS, Christensen O, Calvo E. Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2016 Jul;17(7):883-895. doi: 10.1016/S1470-2045(16)30098-5. Epub 2016 Jun 4. PMID 27269741
- [Background] Ajani JA, D'Amico TA, Bentrem DJ, Chao J, Corvera C, Das P, Denlinger CS, Enzinger PC, Fanta P, Farjah F, Gerdes H, Gibson M, Glasgow RE, Hayman JA, Hochwald S, Hofstetter WL, Ilson DH, Jaroszewski D, Johung KL, Keswani RN, Kleinberg LR, Leong S, Ly QP, Matkowskyj KA, McNamara M, Mulcahy MF, Paluri RK, Park H, Perry KA, Pimiento J, Poultsides GA, Roses R, Strong VE, Wiesner G, Willett CG, Wright CD, McMillian NR, Pluchino LA. Esophageal and Esophagogastric Junction Cancers, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jul 1;17(7):855-883. doi: 10.6004/jnccn.2019.0033. PMID 31319389
- [Background] Yardley DA. nab-Paclitaxel mechanisms of action and delivery. J Control Release. 2013 Sep 28;170(3):365-72. doi: 10.1016/j.jconrel.2013.05.041. Epub 2013 Jun 11. PMID 23770008
- [Background] Paz-Ares L, Vicente D, Tafreshi A, Robinson A, Soto Parra H, Mazieres J, Hermes B, Cicin I, Medgyasszay B, Rodriguez-Cid J, Okamoto I, Lee S, Ramlau R, Vladimirov V, Cheng Y, Deng X, Zhang Y, Bas T, Piperdi B, Halmos B. A Randomized, Placebo-Controlled Trial of Pembrolizumab Plus Chemotherapy in Patients With Metastatic Squamous NSCLC: Protocol-Specified Final Analysis of KEYNOTE-407. J Thorac Oncol. 2020 Oct;15(10):1657-1669. doi: 10.1016/j.jtho.2020.06.015. Epub 2020 Jun 26. PMID 32599071
- [Background] Shui L, Cheng K, Li X, Shui P, Li S, Peng Y, Li J, Guo F, Yi C, Cao D. Durable Response and Good Tolerance to the Triple Combination of Toripalimab, Gemcitabine, and Nab-Paclitaxel in a Patient With Metastatic Pancreatic Ductal Adenocarcinoma. Front Immunol. 2020 Jun 19;11:1127. doi: 10.3389/fimmu.2020.01127. eCollection 2020. PMID 32636837